CLINICAL TRIAL: NCT02243787
Title: A Randomised, Double-blind, Sequential, Ascending Single-dose Study to Evaluate Safety, Tolerability, Biological Activity, and Systemic Exposure of COVA322, a Bispecific TNF-α / IL-17A Antibody Fusion Protein, in Patients With Stable Chronic Moderate-to-severe Plaque Psoriasis
Brief Title: Safety and Tolerability Study of COVA322 in Patients With Stable Chronic Moderate-to-severe Plaque Psoriasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the observed safety profile of COVA322, the sponsor decided to stop the clinical study.
Sponsor: Covagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVA322-SAD-Psoriasis-001
Record Dates: First submitted 2014-09-09; First posted 2014-09-18 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COVA322 (Experimental): single i.v. infusion
  Interventions: Drug: COVA322
- Placebo (Placebo Comparator): single i.v. infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: COVA322
  Arms: COVA322
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is a randomised, double-blind, placebo-controlled, sequential, ascending single-dose, parallel group study to evaluate safety, tolerability, biological activity, and systemic exposure of COVA322 (tumor necrosis factor alpha (TNF-α) / interleukin 17 A (IL-17A) antibody fusion protein) in patients with stable chronic moderate-to-severe plaque psoriasis. Patients will receive ascending single-doses of COVA322 or placebo as a constant-rate i.v. infusion, followed by 12 weeks of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any ethnic origin; women must be of non-childbearing potential
* Aged between 18 to 65 yrs inclusive
* Body weight of ≥ 40 kg and body mass index between 19 - 32 kg/m2 inclusive
* Established diagnosis of moderate to severe plaque psoriasis for at least 6 months prior to screening. The patients must meet all of the following criteria:
* Psoriasis involving ≥ 10% of body surface area
* Requirement of phototherapy or systemic therapy
* Psoriasis Area and Severity Index (PASI) score of ≥ 10
* Physician"s Global Assessment (PGA) score of ≥ 3
* stable disease

Exclusion Criteria:

* History of clinically relevant allergies or idiosyncrasies to COVA322
* Any history of clinically significant drug hypersensitivity following any therapy with a therapeutical biologic, or asthma, urticaria, or other allergic diathesis
* Clinically significant flare of psoriasis during the 12 weeks before randomization
* Current evidence of non-plaque forms of psoriasis
* Currently evidence of drug-induced psoriasis
* Evidence of any serious systemic or local infection within 3 months before screening
* Evidence of subclinical/latent tuberculosis infection
* History or any signs of lymphoproliferative disease, or a known malignancy or a history of malignancy within the previous 5 years
* History or current evidence of autoimmune diseases other than psoriasis
* Women of child-bearing potential
* Recent previous exposure to systemic psoriasis treatments, including anti-TNF-α therapies, immunosuppressive agents such as cyclosporine, mycophenolate, or tacrolimus, and other medications affecting the immune function
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 2.5 times the upper limit of normal (ULN) at screening
* Serum creatinine level ≥ 1.5 times the ULN at screening
* Positive results in any of the virology tests for HIV-Ab, hepatitis C-virus antibody (HCV-Ab) and hepatitis B-virus surface antigen (HBsAg) or hepatitis B core antibody (HBc-Ab)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events as a Measure of Safety and Tolerability | Up to 12 weeks
  The safety and tolerability of COVA322 will be assessed by monitoring the occurrence of local and systemic adverse events or abnormalities as identified by physical examinations, safety lab, vital parameters, ECG and immune response/antibodies to COVA322.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Reich, Prof. Dr. med, Principal Investigator — Sciderm GmbH
Locations (2):
- Germany (2):
  - Charité research organisation, Berlin
  - SCIderm and Clinical Trial Center North, Hamburg

REFERENCES:
- [Derived] Silacci M, Lembke W, Woods R, Attinger-Toller I, Baenziger-Tobler N, Batey S, Santimaria R, von der Bey U, Koenig-Friedrich S, Zha W, Schlereth B, Locher M, Bertschinger J, Grabulovski D. Discovery and characterization of COVA322, a clinical-stage bispecific TNF/IL-17A inhibitor for the treatment of inflammatory diseases. MAbs. 2016;8(1):141-9. doi: 10.1080/19420862.2015.1093266. Epub 2015 Sep 22. PMID 26390837